CLINICAL TRIAL: NCT01615744
Title: Surgical vs. Conservative Treatment of Displaced Intra-articular Calcaneal Fractures: A Prospective, Randomized, Controlled Multicenter Trial
Brief Title: Surgical vs Conservative Treatment of Displaced Intra-articular Calcaneal Fractures: A Prospective RCT
Status: Completed | Type: Observational
Sponsor: Agren, Per-Henrik, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: CalcanealfxRCT
Record Dates: First submitted 2012-06-05; First posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Os Calcis Fracture
Keywords: calcaneal fractures; surgical treatment; conservative treatment; VAS scoring; SF-36; AOFAS; Olerud-Molander score; outcome
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical ORIF calcaneal fx
  Interventions: Procedure: Open Reduction Internal Fixation
- Conservative treatment calcaneal fx
  Interventions: Procedure: Non-surgical management

INTERVENTIONS:
Procedure: Open Reduction Internal Fixation — Lateral approach through extensile lateral incision ( Benirschke), Reduction ( Soeur et Remy) and internal fixation with lateral plating with or without bone graft
  Other Names: Surgery
  Groups: Surgical ORIF calcaneal fx
Procedure: Non-surgical management — Early active exercises and elevation to decrease swelling
  Other Names: No surgery; early movement; decreasing swelling
  Groups: Conservative treatment calcaneal fx

SUMMARY:
Between 1994-98 5 hospitals in Stockholm investigated calcaneal fractures in a randomised study.

82 patients were included and randomized either to non-surgical treatment or surgical management with extensile lateral approach and reduction with Internal fixation (ORIF) The patients were followed and investigated at fixed intervals 2 weeks, 8 weeks, 3 months and 6 months for clinical review. At 1 year and 8-12 years (mean 10 years) post-injury.

Both clinical radiological data were collected and several scores were used. The primary outcomes scores used were SF-36 and VAS score.

The results after 1 year and mean 10 years are presented.

DETAILED DESCRIPTION:
The study was approved by the local ethical committee. Seven trauma orthopaedic surgeons in five hospitals in Stockholm were recruited in this RCT, which was conducted between 1994 and 1998. Patients presented with > 2mm DIACFs verified by axial and coronal computerized tomography (CT) scan were considered for inclusion. Exclusion criteria included peripheral neuro-vascular disease (signs and symptoms of ischemia or neuropathy), open fractures, uncontrolled diabetes mellitus and medical contra-indications to surgery.

All centers used the same study protocol. Demographic data were obtained from the patients, as they deemed eligible to participate in the study. Informed consent was obtained from each patient. Randomization was carried out by sealed opaque envelope to choose surgical vs. conservative treatment.

The surgical treatment was carried out within 2 weeks post-injury when the local soft tissue swelling subsided. Surgery included open reduction using the lateral extensile approach according to Benirschke (ref) and manipulation of the fragments as described by Soeur and Remy (ref) to achieve anatomical reduction, which then was fixed by screws, reconstruction plates or calcaneal plates. Using bone grafts was left to the judgment of the surgeon. Postoperatively, plain X-ray and CT scan were used to evaluate the quality of fracture reduction. Sex week's non-weight bearing was advocated for all patients. Range-of-motion exercises were allowed during this period. Thereafter, the patients had a standardized physiotherapy regimen with full weight bearing.

The conservative treatment included rest, elevation and non-weight bearing. Early range-of-motion exercises were encouraged as tolerated. After 6-8 weeks weight bearing was allowed and shoe modification was provided to those who had hind foot deformities.

No patients were managed with impulse compression therapy.

Patients of both groups were followed-up by treating surgeons at 2 weeks, 8 weeks, 3 months and 6 months for clinical review. At 1 year and 8-12 years (mean 10 years) post-injury, all patients were evaluated by unbiased surgeons who were not involved in the treatment of the patients and they completed the following questionnaires:

1. Primary outcome measures: visual analogue scale (VAS) scoring devised and tested by Hildebrand et al (ref) and a self-administrated general health outcome form (SF-36) for physical and mental health.
2. Secondary outcome measures: VAS at rest and on weight bearing (0-10), the American Orthopaedic Foot & Ankle Society (AOFAS) hindfoot scale and the Olerud-Molander (OM) score.

The investigators divided each group into two subgroups, younger and older than 50 years to determine if the results of the outcome measures at 1 year would differ according to the age of the patients.

During controls, clinical evaluation was carried out to measure the ankle joint and subtalar joint range of motion and the length and width of the hind foot. The contra-lateral non-fractured foot was used for comparison. Shoe problems, the outcome of any eventual postoperative/post-injury complications and workers´ compensation were documented. Radiological follow-up with axial and coronal CT scan was done at the 1 year and 3 years visits.

Statistical analysis The SPSS program version 18.0 for personal computers (Chicago, Illinois) was used for data analysis. The variables of interests were analyzed to determine the differences using bivariate comparisons. The means with standard deviation (SD) were measured. The Mann-Whitney test was used for non-parametric data while two-sample t-test was used for parametric data. A p value of <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with > 2mm DIACFs verified by axial and coronal computerized tomography (CT) scan were considered for inclusion

Exclusion Criteria:

* Peripheral neuro-vascular disease (signs and symptoms of ischemia or neuropathy), open fractures, uncontrolled diabetes mellitus and medical contra-indications to surgery.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between 1994 and 1998. Patients presenting at 5 hospitals in Stockholm after trauma resulting in a fracture with > 2mm Dislocated Intraarticular Calcaneal Fractures (DIACFs) verified by axial and coronal computerized tomography (CT) scan were considered for inclusion
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 1993-12; Primary Completion 1994-01 (Actual); Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
SF-36 | 1 year and 10 years post injury
  The investigators anticipate that there might be a change over time and want to investigate and describe it
VAS-score (calcaneal fractures) /Hildebrand, Buckley | 1 year and 10 years post injury
  The investigators anticipate that there might be a change over time and want to investigate and describe it

SECONDARY OUTCOMES:
VAS of pain at rest and exertion | 2 weeks,6 weeks,12 weeks,1 year, 3 years and 10 years post injury
  The investigators anticipate that there might be a change over time and want to investigate and describe it
AOFAS hindfoot scale | 1 year and 10 years post injury
  The investigators anticipate that there might be a change over time and want to investigate and describe it
Olerud-Molander score | 1 year and 10 years post injury
  The investigators anticipate that there might be a change over time and want to investigate and describe it

CONTACTS AND LOCATIONS:
Overall Officials: Per-Henrik Aagren, MD, Principal Investigator — Consultant Orthopaedic Surgeon
Locations (1):
- Stockholms Fotkirurgklinik, Sophiahemmet, Stockholm, Sweden